CLINICAL TRIAL: NCT00680121
Title: The Effectiveness of Benfotiamine in Reducing Abusive Drinking Among Family History Positive and Negative Alcoholics
Brief Title: High Dose Vitamin B1 to Reduce Abusive Alcohol Use
Acronym: B1AS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Ann Manzardo, PhD, Assistant Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11236
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alcoholism
Keywords: Alcoholism; Benfotiamine; Thiamine
MeSH Terms: conditions — Alcoholism | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Benfotiamine (Experimental): Benfotiamine 600 mg
  Interventions: Drug: Benfotiamine

INTERVENTIONS:
Drug: Benfotiamine — Benfotiamine 600 mg
  Arms: Benfotiamine
Drug: Placebo — Placebo
  Arms: Control Group

SUMMARY:
B1AS tests the hypothesis that increased vitamin B1 (thiamine) intake can repair brain systems damaged by alcohol and help people with alcohol problems control their alcohol use. A strong, man-made form of thiamine (Benfotiamine) is used to increase blood thiamine to much higher levels than can be achieved using normal vitamin supplements. Drinking patterns are examined over 6 months of continued supplement use. Men and women with a recent history of alcohol problems are eligible to participate.

DETAILED DESCRIPTION:
B1AS is a randomized, double-blind placebo-controlled clinical trial of the effectiveness of Benfotiamine at reducing abusive drinking patterns in individuals with recent alcohol problems. Subjects consume 4 tablets of Benfotiamine (600 mg) or placebo daily for 6 months. Monthly follow-ups track alcohol use and alcohol-related problems over the 6 months. Blood tests are also conducted to determine the frequency of an inherited abnormality in thiamine processing that may be related to the risk of developing alcoholism.

ELIGIBILITY:
Inclusion Criteria:

* Problem drinking in the last 30 days

Exclusion Criteria:

* Prolonged abstinence
* Serious medical problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Manzardo, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Manzardo AM, Pendleton T, Poje A, Penick EC, Butler MG. Change in psychiatric symptomatology after benfotiamine treatment in males is related to lifetime alcoholism severity. Drug Alcohol Depend. 2015 Jul 1;152:257-63. doi: 10.1016/j.drugalcdep.2015.03.032. Epub 2015 Apr 8. PMID 25908323

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Placebo; identically matched to Benfotiamine capsules
- Benfotiamine: Benfotiamine 600 mg; 4 capsules taken once daily by mouth for 24 weeks
Period: Overall Study
Arm/Group | Control Group | Benfotiamine
Started | 60 | 60
Completed | 33 | 37
Not Completed | 27 | 23
Not completed — Lost to Follow-up | 27 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Benfotiamine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.7) | 48.1 (6.9) | 47.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 42 | 43 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 43 | 86
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Familial History (FH) of Alcoholism [Number; unit: participants]
  Positive for FH of alcoholism | 51 | 51 | 102
  Negative for FH of alcoholism | 9 | 9 | 18
Alcoholism Severity [Mean (Standard Deviation); unit: scores on a scale] — The alcoholism severity scale measures the severity of a person's dependence to alcohol. The severity is measured from 0 (least severe) to 33 (most severe).
  scores on a scale | 17.9 (6.2) | 16.4 (5.3) | 17.2 (5.8)
Duration of Abuse (years) [Mean (Standard Deviation); unit: years] | 31 (9.8) | 33 (7.6) | 32 (8.8)
Age 1st Drinking (years) [Mean (Standard Deviation); unit: years] | 16 (5.2) | 15 (3.2) | 16 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Alcohol Consumption
Description: measured as standard drinks of alcohol per day (SD/day)
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: alcoholic drinks per day
Arm/Group | Control Group | Benfotiamine
Number analyzed (Participants) | 33 | 37
alcoholic drinks per day | -3.4 (3.6) | -3.0 (4.6)

2. Secondary Outcome: Alcoholism Severity Scale
Description: The alcoholism severity scale measures the severity of a person's dependence to alcohol. The scale ranges from a score of 0 (least severe) to 33 (most severe). The higher the score the worse the dependence.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Benfotiamine
Number analyzed (Participants) | 33 | 37
scores on a scale | 14.0 (5.2) | 10.7 (4.9)

3. Secondary Outcome: Barrett Impulsivity Scale: Total Impulsiveness
Description: Scale measures impulsiveness. It includes 30 items that are scored to yield six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness). Items are scored on a 4 point scale with 1 point equaling rarely/never up to 4 points equaling almost always/always. Total impulsivity score ranges from 30 (least impulsive) to 120 (most impulsive). The higher the score the higher the level of impulsiveness.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Benfotiamine
Number analyzed (Participants) | 33 | 37
scores on a scale | 65.0 (11.4) | 65.4 (9.4)

4. Secondary Outcome: Symptom Checklist-90 (SCL-90): Global Severity Index
Description: The SCL-90 is a brief multidimensional self-report inventory that screens for nine symptoms of psychopathology and provides three global distress indicators. It provides an overview of symptom severity and intensity. The outcome measures psychiatric symptoms using a 30-item scale reported as t-scores relative to a normative population.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Control Group | Benfotiamine
Number analyzed (Participants) | 33 | 37
t-score | 1.02 (0.78) | 1.04 (0.77)

ADVERSE EVENTS:
Arm/Group | Control Group | Benfotiamine
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes